CLINICAL TRIAL: NCT01358929
Title: A Randomized, Placebo-Controlled, Sequential, Multiple-Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MAR701/RO6807952 in Type 2 Diabetic Patients
Brief Title: A Study of RO6807952 in Patients With Diabetes Mellitus Type 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP25742
Record Dates: First submitted 2011-05-18; First posted 2011-05-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO6807952
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to RO6807952
  Arms: 2
Drug: RO6807952 — Escalating subcutaneous dose
  Arms: 1

SUMMARY:
This randomized, placebo-controlled, multiple ascending dose study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of RO6807952. Patients will receive multiple weekly subcutaneous doses of RO6870952. The anticipated time on study treatment is 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 70 years of age, inclusive
* Diagnosis of type 2 diabetes >/=3 months and </=10 years prior to screening
* Fasting plasma glucose >/=110 mg/dL and </=240 mg/dL
* Patients on a stable dose of metformin for at least 2 months prior to screening
* Hemoglobin HbA1c >/=6.5% and </=10.5%
* Body mass index >/=25 kg/m2 and </=42 kg/m2
* Systolic blood pressure <155 mmHg and diastolic blood pressure <95 mmHg

Exclusion Criteria:

* Patients with type 1 diabetes
* History of significant renal and hepatic diseases
* History of metabolic acidosis and diabetic gastroparesis
* History of pancreatitis
* History of coagulation disorders or unexplained excessive bleeding
* History of clinically significant cardiovascular disease or severe symptomatic hypoglycemia within 6 months of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 8 weeks

SECONDARY OUTCOMES:
Blood concentrations of RO6807952 | 8 weeks
Effect of RO6807952 on Hemoglobin HbA1c level | 8 weeks
Effect of RO6807952 on glucose level | 8 weeks
Change in meal tolerance test | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Chula Vista, California
  - Cincinnati, Ohio